CLINICAL TRIAL: NCT01544725
Title: Ketamine-propofol Versus Ketamine Alone for Procedural Sedation in Adults : a Blinded, Randomized Controlled Trial
Brief Title: Ketamine-propofol Versus Ketamine Alone for Procedural Sedation in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-PP-16
Record Dates: First submitted 2012-02-06; First posted 2012-03-06 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Fracture; Dislocation
Keywords: Procedural sedation; Ketamine-propofol; Ketamine
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine-propofol (Experimental)
  Interventions: Drug: Procedural sedation with ketamine-propofol combination
- Ketamine alone (Active Comparator)
  Interventions: Drug: Procedural sedation with ketamine alone

INTERVENTIONS:
Drug: Procedural sedation with ketamine-propofol combination — K= Kétamine P= Propofol RSS= Ramsay Sedation Score
  At t0: 0.5 mg/kg of K (0.1 ml/kg of 5 mg/ml K) followed by 0.5 mg/k of P (0.1 ml/kg of 5 mg/ml P).
  At t0 + 4 min, if needed to obtain an optimal sedation (RSS of 4 or 5): 0.25 mg/kg of K (0.05 ml/kg of 5 mg/ml K) followed by 0.25 mg/kg of P (0.05 ml/kg of 5 mg/ml P).
  At t0 + 8 min, if needed to obtain an optimal sedation (RSS of 4 or 5): 0.25 mg/kg of K (0.05 ml/kg of 5 mg/ml K) followed by 0.25 mg/kg of P (0.05 ml/kg of 5 mg/ml P).
  At t0 + 12 min, if maximal doses have been reached (1 mg/kg of K + 1 mg/kg of P) but the optimal sedation has not been obtained, the procedural sedation will be recorded as a failure in the analysis, and the patient will receive another procedural sedation product (at the discretion of the caregiver).
  Arms: Ketamine-propofol
Drug: Procedural sedation with ketamine alone — K= Ketamine I= Intralipid placebo
  At t0: 1 mg/kg of K (0.1 ml/kg of 10 mg/ml K), followed by 0.1 ml/kg of I (physical placebo of propofol in the other arm).
  At t0 + 4 min, if needed to obtain an optimal sedation (Ramsay Sedation Score of 4 or 5): 0.5 mg/kg of K (0.05 ml/kg of 10 mg/ml K), followed by 0.05 ml/kg of I.
  At t0 + 8 min, if needed to obtain an optimal sedation (Ramsay Sedation Score of 4 or 5): 0.5 mg/kg of K (0.05 ml/kg of 10 mg/ml K), followed by 0.05 ml/kg of I.
  At t0 + 12 min, if maximal doses have been used (2 mg/kg of K) but the optimal sedation has not been obtained, the procedural sedation will be recorded as a failure in the analysis, and the patient will receive another procedural sedation product (at the discretion of the caregiver).
  Arms: Ketamine alone

SUMMARY:
Using Ketamine for procedural sedation in adults is often uncomfortable for emergency physicians because of the significant proportion of patients experimenting recovery agitation. The investigators believe that combining propofol to ketamine, the proportion of recovery agitation will be significantly lowered.

The objectives of this double-blinded, randomized controlled trial are to compare the proportion of recovery agitation in adults receiving procedural sedation with ketamine-propofol versus ketamine alone, and to compare the proportion of other classical procedural sedation side-effects and parameters such as respiratory depression, hypotension, sedation duration, time of recovery, procedural failures, and levels of satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* indication of procedural sedation

Exclusion Criteria:

* allergy to propofol or ketamine
* alcohol or drug intoxication
* altered mental status
* ASA physical status score > 2
* hemodynamic unstability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of recovery agitation | Recovery agitation is noted after procedural sedation for each patient (30 minutes)
  Patient will be followed during the procedural sedation, for an average time of thirty minutes after the first injection

SECONDARY OUTCOMES:
Time from first injection to optimal sedation | Patient will be followed during the procedural sedation, for an average time of thirty minutes after the first injection (30 minutes)
Proportion of respiratory depression | respiratory depression is assessed during procedural sedation for each patient (30 minutes)
  Patient will be followed during the procedural sedation, for an average time of thirty minutes after the first injection
Proportion of arterial hypotension | Hypotension is assessed during procedural sedation for each patient (30 minutes)
  Patient will be followed during the procedural sedation, for an average time of thirty minutes after the first injection
Proportion of vomiting | vomiting is assessed after procedural sedation for each patient (30 minutes)
  Patient will be followed duriong the procedural sedation, for an average time of thirty minutes after the first injection
Recovery time | Recovery time is assessed after procedural sedation for each patient (30 minutes)
  Patient will be followed duriong the procedural sedation, for an average time of thirty minutes after the first injection
Proportion of procedural failures | Procedural failure is noted for each patient if it's happened (30 minutes)
  Patient will be followed duriong the procedural sedation, for an average time of thirty minutes after the first injection
Level of patient's satisfaction | after procedural sedation, patient's satisfaction is recorded (30 minutes)
  Patient will be followed during the procedural sedation, for an average time of thirty minutes after the first injection
Level of care giver's satisfaction | after procedural sedation, care giver's satisfaction is recorded (30 minutes)
  Patient will be followed during the procedural sedation, for an average time of thirty minutes after the first injection

CONTACTS AND LOCATIONS:
Overall Officials: Fabien LEMOEL, MD, Principal Investigator — CHU de Nice, FRANCE; Jacques LEVRAUT, PD, MD, Study Director — CHU de Nice, FRANCE
Locations (1):
- Hôpital St Roch, Nice, France